CLINICAL TRIAL: NCT00586807
Title: Metabolic Response to Infliximab in Pediatric Ulcerative Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Indiana University (Other)
Collaborators: ASPEN Rhoads Research Foundation (Industry)
Responsible Party: Steven J. Steiner, MD, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GCRC 1274; IRB #0503-23
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Ulcerative Colitis; Protein Metabolism; Energy Expenditure
Keywords: Ulcerative colitis; pediatrics; UC; protein metabolism; energy expenditure
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infliximab (Other): Subjects on infliximab
  Interventions: Other: Stable amino acid isotopes

INTERVENTIONS:
Other: Stable amino acid isotopes — Stable amino acid isotopes given per IV, dose based on weight and given over the length of the study visit.

SUMMARY:
The metabolic response to ulcerative colitis, including increased proteolysis and lipolysis and changes in energy expenditure, plays a significant role in the resulting malnutrition from which these patients suffer. Tumor necrosis factor-alpha (TNF-alpha), a pro-inflammatory cytokine, has been found to be elevated in children with ulcerative colitis. TNF-alpha has been incriminated in the mechanism of weight loss in many different chronic diseases, and causes net protein and lipid catabolism. Anti-TNF-alpha antibody (infliximab) has been proven to be an effective therapy for ulcerative colitis.

The purpose of this study is to determine changes in protein and lipid metabolism, as well as resting energy expenditure, before and after therapy with anti-TNF-alpha antibody (infliximab) in children with ulcerative colitis. Performing this study will better define the changes in nutrition status observed in these children following remission of active ulcerative colitis, and potentially lead to changes in medical and nutritional management of these children

ELIGIBILITY:
Inclusion Criteria:

* Male and female children between the ages of six and eighteen years of age
* Endoscopic or histologic evidence of ulcerative colitis
* Active ulcerative colitis determined by primary pediatric gastroenterologist to require anti-tumor necrosis factor-alpha antibody (infliximab) therapy
* Colitis symptom score ≥2
* Screening laboratory tests that meet the following criteria (obtained within 4 weeks of enrollment):

  1. Hemoglobin >8.0 g/dL
  2. White blood cell count >3.5 x 109/L
  3. Neutrophils >1.5 x 109/L
  4. Platelets >100 x 109/L
  5. Aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase levels within 3 times the upper limit of normal.
  6. PPD skin test with skin induration <5 mm.
  7. Signed written consent from the parent/legal guardian and assent from the child to be obtained prior to enrollment.

Exclusion Criteria:

* Female subjects who are pregnant, nursing, or planning pregnancy.
* Concomitant diagnosis or history of congestive heart failure.
* Serious infection in the 3 months prior to enrollment.
* History of prior or current active or latent tuberculosis.
* Immune deficiency syndrome, including documented human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS).
* History of systemic lupus erythematosus.
* A transplanted organ.
* Known malignancy or history of malignancy within 5 years of enrollment.
* History of demyelinating disease.
* History of substance abuse.
* History of diabetes mellitus.
* Poor tolerability of venipuncture or lack of venous access during the study period.
* A live virus vaccination within 3 months of enrollment.
* Prior history of infliximab infusion or any other therapeutic agent targeted at reducing tumor necrosis factor-alpha (TNF-alpha).
* Hypersensitivity to any murine proteins or other component of the product.
* Inability to comply with study procedures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Measure protein kinetics and balance in response to anti-TNF-alpha therapy in children with steroid-resistant ulcerative colitis, during both the fasting state and parenteral nutrition infusion. | Week 0 and 2

SECONDARY OUTCOMES:
2. Measure energy expenditure by indirect calorimetry in response to anti-TNF-alpha therapy in children with steroid-resistant ulcerative colitis, during both the fasting state and parenteral nutrition infusion. | Week 0 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Steiner, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University- Riley Hospital for Children, Indianapolis, Indiana, United States